CLINICAL TRIAL: NCT07399899
Title: A Phase 1, Dose-Escalating Crossover, Pharmacokinetic/Pharmacodynamic Study, Assessing the Safety and Pharmacokinetics of NBX-100 in Healthy Adult Participants
Brief Title: Dose-Finding Study of NBX-100 in Healthy Adult Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neurala Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB-2025 P1 001
Record Dates: First submitted 2025-11-16; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: Multiple Ascending Dose (MAD) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NBX-100 (Experimental): NBX-100 oral capsules
  Interventions: Drug: NBX-100

INTERVENTIONS:
Drug: NBX-100 — NBX-100 comprises of a tryptamine and two other MAOI compounds

SUMMARY:
NB-2025 P1 001 is a Phase Ib study that will investigate the pharmacokinetics, pharmacodynamics, safety, tolerability, psychological effects of escalating doses of NBX-100 in healthy volunteers.

A 28-day screening period is followed by a preparation visit with psychologist in Week 1. From Week 2 to Week 5, participants will receive a once weekly dose of study treatment, receiving four doses in total. Participants will attend a follow-up visit each day immediately after each dosing day. In Week 6, participants will attend an integration visit with a psychologist, and in Week 10, participants will attend an end-of-study follow-up visit.

Participants will have safety, psychological, PK, PD, and pharmacogenomic assessments.

DETAILED DESCRIPTION:
NB-2025 P1 001 is a Phase I, single-centre study that will investigate the pharmacokinetics, pharmacodynamics, safety, tolerability, psychological effects of escalating doses of NBX-100 in healthy volunteers.

A total of eight (8) participants will be enrolled overall, split into two cohorts of four (4) participants. This split into two cohorts is for logistical purposes, as there is a maximum of four participants allowable per cohort in the facility to provide sufficient safety oversight. Participants will attend the clinic as part of their cohort for individual dosing sessions, with dosing to be performed in separate dosing rooms. Doses for each participant will be staggered per PI discretion, and each participant may be separated into individual dosing rooms to avoid social contagion effects. Doses will be the equivalent of 10, 40, 80 or up to 120 mg of a tryptamine, ascending from 10 mg at Dose 1 to at most 120 mg at Dose 4. The tryptamine will be given in combination with an MAOI-a combination.

Following a 28-day Screening period (Day -28 to Day -1), participants will attend a preparation session in Week 1, the week prior the first dosing session, with a clinical psychologist, and be provided with supportive preparation material. In the Week 2 to 5 visits, participants will attend a one-on-one session with a clinical psychologist the night before each dosing day, at the facility, then stay overnight. On each dosing day, participants will be administered a single dose of study treatment (NBX-100 capsules) according to the dosing schedule. Participants will remain at the facility for monitoring and assessment. At the end of the day, after medical assessment and sign off from the Investigator, participants are to be picked up by a nominated person for transport. An overnight stay after the dose is optional, if requested by the study team or the participant. In the event of an adverse event the medical and psychologist team will either have the participant stay overnight, or offer appropriate management strategy if the participant declines to stay. Participants are to return the following day for follow-up assessments. In Week 6, participants are to attend an Integration session with a clinical psychologist. The End-of-Study/Follow-up visit will occur in Week 10.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 21-50 years of age (inclusive).
2. Able and willing to provide written informed consent prior to the performance of any study-specific procedures.
3. Able and willing to comply with all scheduled visits, study treatment, laboratory tests, lifestyle considerations, and other study procedures.
4. Has a nominated person to collect them from the study site in the afternoon/evening of each dosing day and then drive them home.
5. Medically and psychiatrically healthy as judged by the Principal Investigator or delegate based on medical history, physical examination, vital signs, laboratory tests, and 12-lead ECG.
6. At least 2 prior ayahuasca experiences within the previous 5 years relative to Screening, but none within the last month
7. Have a Body Mass Index (BMI) between 18.0 and 32.0 kg/m2 (inclusive) and a body weight ≥50 kg.
8. Female participants of childbearing potential must have a negative serum pregnancy test at Screening, and a negative urine pregnancy test at Day 1.
9. Female participants of childbearing potential must be willing to use two highly-effective methods of contraception simultaneously from date of consent, and for 30 days after the last dose of study intervention, and must not breastfeed for the same period of time. They are not to donate any ova from the date of first dose and for 30 days after the last dose of study intervention. Approved contraception methods are:

   * The use of TWO of the following:

     * The use of a barrier method of contraception (i.e., a condom or diaphragm);
     * Established use of oral, injected or implanted hormonal methods of contraception; or
     * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * Or, either of the below:

     * Sterilised male partner; or
     * Abstinence from penile-vaginal intercourse.
10. Women who are not of child-bearing potential may be enrolled and are defined as women who:

    * have been surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, and/or tubal ligation); or
    * are post-menopausal, as defined by amenorrhoea for at least 12 consecutive months (and not induced by medical conditions such as anorexia nervosa and not taking medications that induced the amenorrhea, e.g., oral contraceptives, hormones, gonadotropin releasing hormones, anti-estrogens, selective estrogen receptor modulators, or chemotherapy).
11. Male participants are eligible if they have had a documented vasectomy or are willing to use two highly-effective methods of contraception simultaneously from date of consent, and up to 10 weeks after the last dose of study intervention and must not donate sperm from the date of first dose to 10 weeks after the last dose of study intervention. Approved contraception methods are:

    * The use of TWO of the following:

      * The use of a barrier method of contraception (i.e., a condom or diaphragm);
      * Established use of oral, injected or implanted hormonal methods of contraception; or
      * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * Or, either of the below:

      * Surgically sterilised female partner; or
      * Abstinence from penile-vaginal intercourse.

Exclusion Criteria:

1. History of psychosis: past or present diagnosis of bipolar disorder type 1 or type 2, schizophrenia, schizoaffective disorder, major depressive disorder, dysthymia, anxiety disorders, and post-traumatic stress disorder.
2. Family history of psychosis: past or present diagnosis of bipolar disorder type 1 in first degree relative,
3. Family history of psychosis: past or present diagnosis of schizophrenia or schizoaffective disorder in first or second degree relative.
4. Current suicidality, or history of suicide attempt.
5. Cannot tolerate venipuncture.
6. Is not a good candidate for cannulation and/or multiple PK blood draws, as determined by the Principal Investigator or delegate.
7. Has a known or suspected hypersensitivity or allergic reaction to any of the ingredients of the study medication.
8. High-risk alcohol use (defined as more than 10 standard drinks per week on average over the last 3 months) or history of alcohol abuse in the last 2 years.
9. Has taken prescription medication within 30 days prior to first dose of study medication. A washout can be employed.
10. Has taken over-the-counter drugs, including dietary supplements, herbal supplements and traditional medicines within 14 days prior to first dose of study medication. A washout can be employed. Permitted medications for use during the study (but not on the treatment day), include the irregular use of non-opiate analgesics, e.g., paracetamol; the oral contraceptive pill; general nutraceuticals, e.g., vitamins.
11. Regular smoking (no more than 5 cigarettes or equivalent nicotine products including patches and vapes per week on average over the last 6 months) or any other current substance use disorder (alcohol, amphetamine, cocaine, opiates).
12. Positive urine drug screen for substances listed on a drug abuse panel (e.g., methamphetamines, cocaine, cannabinoid/THC, phencyclidine, benzodiazepines, amphetamines, methadone, opiates, tricyclic antidepressants, barbiturates, or cotinine). Urine drug screen may be repeated once at the discretion of the Principal Investigator or delegate.
13. Serious medical condition including insulin-dependent diabetes or history of hypoglycaemia, seizure disorder or epilepsy, coronary artery disease, heart failure, cancer, history of cerebrovascular event, uncontrolled or medicated adult asthma, hyperthyroidism, cardiovascular conditions: uncontrolled hypertension, angina, TIA, stroke, peripheral or pulmonary vascular disease.
14. Impaired liver function (ALT or AST > 1.5 × upper limit of normal).
15. Renal function issues (eGFR < 60 mL/min/1.73m2, by CKD-EPI equation).
16. Persistently elevated blood pressure (systolic blood pressure above 160 mmHg or diastolic blood pressure above 95 mmHg).
17. Clinically significant ECG abnormality (including QTcF abnormalities, ≤450 for males and ≤470 for females) at Screening, as determined by the Principal Investigator or delegate.
18. Abnormal hematology or blood chemistry test result(s) deemed clinically significant at Screening or Week 1, as determined by the Principal Investigator or delegate.
19. Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV)-1 or HIV-2 antibody at Screening.
20. Has participated in any clinical trial or received an investigational product within 3 months or 5 half-lives of the product (whichever is longer) prior to Screening.
21. Has donated blood or had non physiological blood loss of more than 200 mL within 3 months prior to Screening.
22. Has an active infection in the 7 days prior to first dose of study medication) that may interfere with study assessments. Inclusion to be assessed and confirmed by the Principal Investigator or delegate.
23. Has any condition which could confound the results of the study, interfere with participation in the study or increase the risks of study participation, in the opinion of the Principal Investigator or delegate.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (last) | Up to 24 hours post-dose
  AUC0-last across 11 timepoints
Area under the plasma concentration versus time curve (zero to infinity) | Up to 24 hours post-dose
  AUC0-inf across 11 timepoints
Peak plasma concentration | Up to 24 hours post-dose
  Cmax across 11 timepoints
Time to peak drug concentration | Up to 24 hours post-dose
  Tmax across 11 timepoints
Elimination half-life | Up to 24 hours post-dose
  t1/2 across 11 timepoints
Apparent drug clearance | Up to 24 hours post-dose
  C/F across 11 timepoints

SECONDARY OUTCOMES:
Assessment of AEs | Baseline, Day 1, Day 2, Day 5, Day 35
  Number of participants with treatment-emergent adverse events, categorized by system organ class
Tolerability of NBX-100 | Day 1, Day 2, Day 5, Day 35
  Number of participants experiencing adverse events related to study drug
Use of rescue medications | Day 1, Day 2
  type of medication
Change from baseline in diastolic blood pressure | Baseline, Day 1, Day 2, Day 7, Day 35
  Mean change from baseline in diastolic blood pressure (mmHg)
Clinical laboratory blood tests | Baseline, Day 1, Day 35
  Number of participants with abnormal laboratory tests results
Psychological distress scale | Baseline, Day 2, Day 7, Day 35
  visual analogue scale 1-100 (higher or lower, whereby a higher score indicates greater psychological distress)
Drug Liking Scale | Day 1, Day 2, Day 7, Day 35
  visual analogue scale 1-100 (higher or lower; whereby a higher score indicates a greater liking for the drug)
Columbia-Suicide Severity Rating Scale | Baseline, Day 1, Day 7, Day 35
  Change in suicidal ideation severity level as assessed by the Columbia-Suicide Severity Rating Scale (severity levels 1-5)
Pulse rate change | Baseline, Day 1, Day 2, Day 7, Day 35
  Change from baseline in pulse rate (beats per minute)
Change from baseline in systolic blood pressure | Baseline, Day 1, Day 2, Day 7, Day 35
  Mean change from baseline in systolic blood pressure (mmHg)

OTHER OUTCOMES:
Self-reported subjective psychedelic intensity rating, by dose level | Day 1, Day 2
  Mean self-reported subjective psychedelic intensity rating (1-10), by dose level, measured at multiple points on Day 1 and Day 2 of each Treatment Period
Regensburg Insomnia Scale | Baseline, Day 5, Day 35
  Assessment of insomnia 0-40 (higher score level equating to poorer sleep)
Activity counts or Electrodermal Activity (EDA) level by dose level | Baseline, Day 1, Day 2
  Mean change from baseline in electrodermal activity (EDA), measured in microsiemens (µS), by dose level
CYP2D6 Metabolizer Phenotype | Baseline
  Assessment of participant CYP2D6 alleles to determine metabolizer phenotype: Poor metabolizer; Intermediate metabolizer; Normal/Extensive metabolizer; Ultrarapid metabolizer
Kessler-10 scale | Baseline, Day 2, Day 5, Day 35
  Assessment of mood 0-40 (higher score level equating to lower perceived mood)
Generalised Self-Efficacy Scale | Baseline, Day 2, Day 5, Day 35
  Assessment of perceived self-efficacy 10-40 (higher score level equating to higher levels of self-efficacy)
Total 5D-ASC (5-Dimension Altered States of Consciousness Scale) and dimensions, by dose level | Day 2
  5D-ASC Dimensions (0-100): Experience of Unity, Spiritual Experience, Blissful State, Insightfulness, Disembodiment, Impaired control and cognition, Anxiety, Complex Imagery, Elementary Imagery, AudioVisual Synesthesia, Changed Meaning of Percepts, by dose level
Total MEQ30 (Revised 30-item Mystical Experience Questionnaire) and factors, by dose level | Day 2
  Mean total MEQ30 (0-100) and individual dimensions of Mystical, Positive Mood, Transcendence of Time and Space, and Ineffability, by dose level, with a higher score indicating a stronger mystical experience
Total Short-Index of Mystical Experience (SIME), by dose level | Day 1
  Mean total SIME (0-100) by dose level, measured on Day 1 of each Treatment Period, with a higher score indicating a stronger mystical experience
Persisting Effects Questionnaire summary items by dose level | Day 5
  Mean Persisting Effects Questionnaire 0-100 (how personally: meaningful, spirituality significant, psychological challenging, insightful, wellbeing enhancing) by dose level, measured at Day 5 of each Treatment Period and End-of-Study Visit

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Proprietary company information